CLINICAL TRIAL: NCT03634969
Title: A Phase 1, Open-Label Study to Evaluate the Pharmacokinetics, Safety and Tolerability of BMS-986224 in Participants With Varying Degrees of Renal Function
Brief Title: An Investigational Study to Evaluate Experimental Medication BMS-986224 in Renally Impaired Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CV016-010
Record Dates: First submitted 2018-08-15; First posted 2018-08-17 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Cardiac Failure; Myocardial Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Normal Renal Function (Experimental)
  Interventions: Drug: BMS-986224
- Mild Renal Impairment (Experimental)
  Interventions: Drug: BMS-986224
- Moderate Renal Impairment (Experimental)
  Interventions: Drug: BMS-986224
- Severe Renal Impairment (Experimental)
  Interventions: Drug: BMS-986224
- End-Stage Renal Disease (ESRD) (Experimental): ESRD participants and are on chronic hemodialysis
  Interventions: Drug: BMS-986224

INTERVENTIONS:
Drug: BMS-986224 — Specified dose on specified days

SUMMARY:
The purpose of this study is to investigate the experimental medication BMS-986224 in participants with varying levels of renal function.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* BMI ≥18 and ≤ 35kg/m2
* Systolic blood pressure >100 mmHg

Exclusion Criteria:

* Women of childbearing potential or women who are currently pregnant
* Clinically relevant abnormal medical history, abnormal findings on physical examination, vital signs, ECG, or laboratory tests at screening that the investigator judges as likely to interfere with the objectives of the trial or the safety of the volunteer
* Current or recent (within 3 months of study treatment administration) gastrointestinal disease that could affect absorption

Other protocol defined inclusion/exclusion criteria could apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of BMS-986224 | Up to 11 days
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration [AUC(0-T)] of BMS-986224 | Up to 11 days
Area under the plasma concentration-time curve from time zero to 72 h post dose [AUC(0-72)] of BMS-986224 | Up to 11 days
Area under the plasma concentration-time curve from time zero extrapolated to infinite time [AUC(INF)] of BMS-986224 | Up to 11 days
Time of maximum observed plasma concentration (Tmax) of BMS-986224 | Up to 11 days
Terminal elimination half-life (T-HALF) of BMS-986224 derived from plasma concentration | Up to 11 days
Fraction of unbound drug in plasma (fu) of BMS-986224 | Up to 11 days
Apparent oral clearance (CL/F) of BMS-986224 derived from plasma concentration | Up to 11 days
Apparent volume of distribution (Vz/F) of BMS-986224 derived from plasma concentration | Up to 11 days
Cumulative amount of unchanged drug excreted into the urine at a given time (Aet) of BMS-986224 | 7 days
  Part 1 only
Fraction of dose excreted in urine (Fe%) of BMS-986224 | 7 days
  Part 1 only
Renal clearance of BMS-986224 derived from urine concentration | 7 days
  Part 1 only

SECONDARY OUTCOMES:
Incidence of nonserious adverse events (AE), serious adverse events (SAE), and AE leading to discontinuation | Up to 41 days
Maximum observed plasma concentration (Cmax) of metabolite | Up to 11 days
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration [AUC(0-T)] of metabolite | Up to 11 days
Area under the plasma concentration-time curve from time zero to 72 h post dose [AUC(0-72)] of metabolite | Up to 11 days
Area under the plasma concentration-time curve from time zero extrapolated to infinite time [AUC(INF)] of metabolite | Up to 11 days
Time of maximum observed plasma concentration (Tmax) of metabolite | Up to 11 days
Terminal elimination half-life (T-HALF) of metabolite derived from plasma concentration | Up to 11 days
Metabolite-to-parent (MR) ratio for cMax | Up to 11 days
Metabolite-to-parent (MR) ratio for AUC(0-T) | Up to 11 days
Metabolite-to-parent (MR) ratio for AUC(0-72) | Up to 11 days
Metabolite-to-parent (MR) ratio for AUC(INF) | Up to 11 days
Number of clinically significant changes in vital signs, ECGs, physical examinations, or clinical laboratory tests | Up to 11 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- United States (3):
  - Clinical Pharmacology of Miami, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Prism Research, Saint Paul, Minnesota

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm